CLINICAL TRIAL: NCT06344637
Title: Effects of Cervical Lidocaine Spray on Pain Relief During Manual Vacuum Aspiration : A Randomized Controlled Trial
Brief Title: Effects of Cervical Lidocaine Spray on Pain Relief During Manual Vacuum Aspiration
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UdonThani Hospital (Other Government)
Responsible Party: Principal Investigator, Metha Songthamwat, Principal investigator, UdonThani Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2566/081 I
Record Dates: First submitted 2024-02-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Pain, Procedural; Lidocaine; Obstetric Surgical Procedures
Keywords: manual vacuum aspiration; pain score; Lidocaine spray
MeSH Terms: conditions — Pain, Procedural | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10% lidocaine spray without adrenaline (Experimental): 4 puffs of 10% lidocaine spray without adrenaline apply on cervical os before manual vacuum aspiration
  Interventions: Drug: 10 % lidocaine spray without adrenaline
- Placebo (Placebo Comparator): 4 puffs of normal saline apply on cervical os before manual vacuum aspiration
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 10 % lidocaine spray without adrenaline — Pateint with indication for manual vacuum aspiration aged between 20-60 years will received a standard injection of pethidine along with 1% lidocaine spray without adrenaline on cervical os to compare pain scores with placebo. Along with measuring side effects immediately and 30 minutes after receiving 1% lidocaine without adrenaline.
  Other Names: 10% Xylocaine spray
  Arms: 10% lidocaine spray without adrenaline
Other: Placebo — 4 puffs of normal saline apply on cervical os before manual vacuum aspiration
  Arms: Placebo

SUMMARY:
This randomized control trial aim to evaluate the effectiveness of local lidocaine spray application to the cervix on the reducing of pain score during the manual vacuum aspiration

DETAILED DESCRIPTION:
This is a double blinded, placebo controlled study which compose of two arms. The treatment group is the local lidocaine spray application to the cervix with the intravenous opioid. The control group is the the intravenous opioid with the placebo (normal saline) before the manual vacuum aspiration. The outcome is to compare the visual analog pain score during and after procedure.

ELIGIBILITY:
Inclusion Criteria:

* female ageed 20 years to 60 years who have an indication for manual vacuum adpiration under intraveneous analgesia

Exclusion Criteria:

* patient with allergic to lidocaine or history of allergic to lidocaine
* patient with reproductive and urinary infection
* patient with abnormal vital sign
* patient with abnormal kidney and liver function test

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
pain score during manual vauum aspiration | during surgery
  The pain score using visual analog scale is used to assess the pain score during the manual vacuum aspiration during procedure (score 0-10), the 0 score is no pain and the 10 score is the maximum pain
pain score after manual vauum aspiration | at 30 minutes postoperative
  The pain score using visual analog scale is used to assess the pain score after the procedure (score 0-10) the 0 score is no pain and the 10 score is the maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: PATTARIKAN MANAYING, Principal Investigator — UdonThani Hospital
Locations (1):
- UdonThani Hospital, Udon Thani, UdonThani, Thailand

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT06344637/Prot_SAP_000.pdf